CLINICAL TRIAL: NCT06661265
Title: Predictors of Acute Toxicity and Flap Failure After Adjuvant Treatment for Locally Advanced Head and Neck Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Aurora Mirabile, Medical Oncologist, IRCCS San Raffaele
Other Study IDs: Lembi
Record Dates: First submitted 2024-10-23; First posted 2024-10-28 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer
Keywords: flap reconstructions; flaps; Head and Neck cancer; toxicities; adjuvant chemoradiation
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Surgical Flaps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- SCCHN patients undergoing to upfront surgery with flap reconstruction followed by adjuvant treatment: Head and Neck cancer patients undergoing to upfront surgery with flap reconstruction followed by radiotherapy or chemioradiotherapy at San Raffaele Hospital between December 2017-December 2022.
  Interventions: Procedure: adjuvant tomotherapy +- chemotherapy after the reconstructive surgery with flaps

INTERVENTIONS:
Procedure: adjuvant tomotherapy +- chemotherapy after the reconstructive surgery with flaps — adjuvant treatment in locally-advanced head and neck cancers submitted to upfront surgery with flap reconstruction, evaluation of toxicity and flap status performed at San Raffaele Hospital between December 2017-December 2022.

SUMMARY:
Head and Neck cancer treatment may have significant functional consequences. Decisions about treatment are usually hard to make, as they must strike a balance between efficacy of the treatment and likelihood of survival. Reconstructive surgery with flaps plays a key role in the head and neck cancer resection in order to achieve local control, but often leaves a large, disfiguring composite defect that not only compromises the patient's functional and aesthetic outcome, but also significantly affects quality of life.

Adjuvant treatment, including post operative Radiation Therapy (poRT) and chemotherapy, is crucial in improving locoregional control and survival in locally-advanced cases and the flaps are usually included in radiotherapy fields.

Fourthysix patients undergoing to reconstructive surgery followed by radiation or chemioradiation between Decembre 2017 to December 2022 at San Raffaele Hospital will be enrolled in this study. The first aim of the study is to understand potential predictors of the occurrence of overall acute toxicity following adjuvant treatment in locally-advanced head and neck cancers submitted to upfront surgery with flap reconstruction. By analyzing patient data and treatment variables, the study aims at identifying factors that may influence the incidence and severity of acute treatment-related toxicities, such as mucositis, dysphagia, xerostomia and dermatitis.

The second aim of the study is to evaluate whether the same variables may influence the viability and integrity of the flap at the end of the adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced head and neck cancer squamocellular carcinoma
* treated with post operative radiotherapy +/- chemotherapy
* surgical resected with flap reconstruction

Exclusion Criteria:

* salvage surgery after primary relapse
* previously irradiated
* recurrent/metastatic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally-advanced head and neck cancers' patients undergone adjuvant treatment after upfront surgery with flap reconstruction
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of acute toxicity post adjuvant treatment of tomotherapy +- chemotherapy after the reconstructive surgery with flaps | End of treatment course (up to 6 months)
  Acute toxicity post adjuvant treatment of tomotherapy +- chemotherapy after the reconstructive surgery with flaps will be measured according to Standard Common Criteria for Adverse Events (CTCAE) v5, thus graded as low (G0-1) versus relevant (G2 or more).

SECONDARY OUTCOMES:
Evaluation of the flap status at the end of the adjuvant treatment course of tomotherapy +- chemotherapy after the reconstructive surgery with flaps | End of treatment course (up to 6 months)
  Flap status will be categorized as Healthy (a successful reconstruction with good blood supply, intact tissue viability, and absence of complications) versus Damaged (complications such as partial or total flap loss, flap necrosis, and wound dehiscence, managed with either conservative procedures or revision surgery).